CLINICAL TRIAL: NCT02969720
Title: Double Blind, Randomized, Phase III, Parallel, Placebo-controled Study to Evaluate Therapeutic Efficacy of 2 Grams Phytosterols Daily Supplemention on Patients With Metabolic Syndrome
Brief Title: Therapeutic Efficacy of Phytosterols on Metabolic Syndrome
Acronym: FESIME
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universidad de los Andes, Chile (Other)
Responsible Party: Principal Investigator, Yasna Palmeiro-Silva, Asistant Professor, Universidad de los Andes, Chile
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: FESIME-016
Record Dates: First submitted 2016-11-17; First posted 2016-11-21 (Estimated); Last update posted 2020-03-17 (Actual); Status verified 2020-03

CONDITIONS: Metabolic Syndrome x
MeSH Terms: conditions — Metabolic Syndrome | interventions — Phytosterols; titanium dioxide

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Phytosterol (Experimental): Daily consumption of 2 grams (8 ml) nano-phytosterols per 180 days.
  Interventions: Dietary Supplement: Phytosterols
- Placebo (Placebo Comparator): Daily consumption of 8 ml of a solution with Titanium Dioxide per 180 days.
  Interventions: Dietary Supplement: Titanium Dioxide

INTERVENTIONS:
Dietary Supplement: Phytosterols — Oral daily consumption of 2 grams of phytosterols (8 ml) per 180 days.
  Other Names: Cardiosmile
  Arms: Phytosterol
Dietary Supplement: Titanium Dioxide — Oral daily consumption of Titanium Dioxide (8 ml) per 180 days.
  Arms: Placebo

SUMMARY:
The objective is to evaluate therapeutic efficacy of 2 grams nano-phytosterols daily supplemention on diagnosis criteria of metabolic syndrome.

ELIGIBILITY:
Inclusion Criteria:

* Informed consent written
* Available subjects to follow-up visits
* Subjects with diagnoses of metabolic syndrome 5 years ago or with current diagnoses criteria
* Subjects with health visits ongoing
* Subjects with arterial hypertension under control.
* Subjects with mellitus diabetes under control.

Exclusion Criteria:

* Subjects with alcoholism history.
* Subjects with history of sitosterolemia.
* Subjects with familiar hypercholesterolemia
* Subjects who are consuming phytosterols
* Pregnancy women
* Breastfeeding period women
* Subjects with personal history of: acute miocardical infarction, stroke, hypertensive emergency, acute or chronic diabetes descompensation

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 220 (Actual)
Dates: Start 2018-01-08 (Actual); Primary Completion 2018-11-27 (Actual); Study Completion 2018-11-27 (Actual)

PRIMARY OUTCOMES:
Difference of proportion between study groups in the proportion of metabolic syndrome from baseline and the last visit (180 days). | 180 days

CONTACTS AND LOCATIONS:
Locations (1):
- Universidad de Los Andes, Santiago, Chile

IPD SHARING:
Plan to Share IPD: Undecided
PI will share IPD after doing all possible publications.

REFERENCES:
- [Derived] Palmeiro-Silva YK, Aravena RI, Ossio L, Parro Fluxa J. Effects of Daily Consumption of an Aqueous Dispersion of Free-Phytosterols Nanoparticles on Individuals with Metabolic Syndrome: A Randomised, Double-Blind, Placebo-Controlled Clinical Trial. Nutrients. 2020 Aug 10;12(8):2392. doi: 10.3390/nu12082392. PMID 32785036